CLINICAL TRIAL: NCT05624905
Title: Prospective Registry for Identifying Long-term Prognosis in Patients Who Underwent Coronary Angiography and Percutaneous Coronary Intervention for Coronary Artery Disease
Brief Title: Prospective Pecutaneous Coronary Intervention Registry
Acronym: SMC-PCI
Status: Recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Joo-Yong Hahn, Professor, Samsung Medical Center
Other Study IDs: SMC-PCI
Record Dates: First submitted 2022-11-15; First posted 2022-11-22 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Coronary Artery Disease; Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PCI group: All consecutive patients with coronary artery disease who underwent percutaneous coronary intervention
  Interventions: Procedure: Percutaneous coronary intervention

INTERVENTIONS:
Procedure: Percutaneous coronary intervention — Percutaneous Coronary Intervention Procedure

SUMMARY:
Coronary artery disease is the most important cause of death worldwide. Treatment option for coronary artery disease is medical treatment, percutaneous coronary intervention, or coronary artery bypass surgery. Among them, the field of percutaneous coronary intervention is rapidly developing with regard to the improvement of devices, techniques, or medical treatment, leading to reduce mortality or morbidity. Until now, numerous previous studies related to the risk factors of coronary artery disease and the prognosis of patients have been conducted. However, the field of percutaneous coronary intervention is rapidly evolving, and treatment strategies are constantly being updated. Therefore, the current study sought to identify the long-term prognosis and related risk factors of patients with coronary artery disease who underwent percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

* patients who have undergone or are scheduled to undergo coronary angiography and percutaneous coronary intervention.

Exclusion Criteria:

* patients who did not consent to the research

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients who underwent coronary angiography adn percutaneous coronary intervention
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2016-03-20 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Rates of Cardiac death or Target-vessel myocardial infarction | up to 10 years
  A composite of cardiac death or target vessel myocardial infarction
Rates of Major adverse cardiac and cerebrovascular event | up to 10 years
  A composite of all-cause death, myocardial infarction, cerebrovascular accident, or repeat revascularization

SECONDARY OUTCOMES:
Rates of all-cause death | up to 10 years
  Death from any cause
Rates of cardiac death | up to 10 years
  Death from cardiac cause
Rates of myocardial infarction | up to 10 years
  Any myocardial infarction
Rates of target-vessel myocardial infarction | up to 10 years
  target-vessel myocardial infarction
Rates of target lesion revascularization | up to 10 years
  target lesion revascularization
Rates of target vessel revascularization | up to 10 years
  target vessel revascularization
Rates of cerebrovascular accident | up to 10 years
  ischemic or hemorrhagic stroke
Rates of stent thrombosis | up to 10 years
  definite or probable stent thrombosis

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choi KH, Lee SY, Song YB, Park TK, Lee JM, Yang JH, Choi JH, Choi SH, Gwon HC, Hahn JY. Prognostic Impact of Operator Experience and IVUS Guidance on Long-Term Clinical Outcomes After Complex PCI. JACC Cardiovasc Interv. 2023 Jul 24;16(14):1746-1758. doi: 10.1016/j.jcin.2023.04.022. PMID 37495350